CLINICAL TRIAL: NCT03879486
Title: A Randomized Controlled Trial to Investigate the Infectious Outcomes of Intrarectal Povidone-iodine Cleansing Plus Formalin Disinfection of Needle Tip During Transrectal Ultrasound Guided Prostate Biopsy
Brief Title: Infectious Outcomes of Povidone-iodine Rectal Cleansing Plus Formalin Disinfection of Needle During Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Transplante Doutor Euryclides de Jesus Zerbini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BIOPSY1
Record Dates: First submitted 2018-11-01; First posted 2019-03-18 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Prostate Biopsy; Prostatitis
MeSH Terms: conditions — Prostatic Neoplasms; Prostatitis

STUDY DESIGN:
Intervention Model Description: Prospective controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVPI intervention (Experimental): rectal cleansing and disinfection of the needle tip at transrectal ultrasound guided prostate biopsy
  Interventions: Other: Intrarectal povidone-iodine cleansing plus formalin disinfection of needle tip during transrectal ultrasound guided prostate biopsy
- Control arm (No Intervention): controls at transrectal ultrasound guided prostate biopsy

INTERVENTIONS:
Other: Intrarectal povidone-iodine cleansing plus formalin disinfection of needle tip during transrectal ultrasound guided prostate biopsy — The examiner will use a gauze soaked and saturated with iodopovidone and perform a mechanical friction motion on the anterior wall of the rectum, at least 5 times from one margin to another of the prostate laterally-laterally. A period of two (2) minutes shall be waited from the prophylactic cleaning of the rectum to the beginning of the biopsy. The examiner will use a technique of disinfecting the 10% formaldehyde biopsy needle without manual contact by soaking the distal 3 cm of the needle directly into a vial containing the bactericidal solution between obtaining the different fragments. An individual bottle will be used for each patient
  Arms: PVPI intervention

SUMMARY:
The main purpose of this study is to compare the infectious outcomes of intrarectal povidone-iodine cleansing plus formalin disinfection of needle tip during transrectal ultrasound guided prostate biopsy. The secondary objective is to evaluate predictive factors of infectious complications after prostate biopsy. Data will be prospectively collected from patients who will undergo prostate biopsy in a single high volume urology center. The patients will be randomized to two different groups: group A - rectal cleansing and disinfection of the needle tip vs group B - controls.

DETAILED DESCRIPTION:
Prostate cancer is the most common neoplasm of solid organs in Brazil. Definitive diagnosis of the tumor is established through prostate biopsy, indicated in patients with elevated levels of PSA or suspicious rectal examination. The ultrasound or MRI-guided prostate biopsy is mostly performed through the transrectal route worldwide. Although it is a relatively safe procedure, transrectal prostate biopsy (TRUSB) can present several complications, such bleeding, acute urinary retention or infection. Infectious complications are an important concern for the urologist and have different presentation, ranging from isolated fever to severe sepsis. Antibiotic prophylaxis is an effective widely used practice, however, due to increasing rates of bacterial resistance, there is a growing trend in the incidence of infectious complications after TRUSB. Therefore, alternative strategies to decrease infections rates following biopsies are welcome. Our aim was to compare the infectious complications of intrarectal povidone-iodine cleansing associated to formalin disinfection of biopsy needle tip at prostate biopsy.

A prospective controlled study will be conducted enrolling 1152 consecutive prostate biopsies in a single center high volume urology Brazilian Public Hospital. The patients will be randomized at a 1: 1 ratio for two different groups: group A - rectal cleansing and disinfection of the needle tip vs. Group B - controls at transrectal ultrasound guided prostate biopsy. Patients will obtain a urine culture 48 hours after biopsy and complete a telephone interview 7 days after undergoing the procedure. The primary endpoint will be the rate of infectious complications, defined as 1 or more of the following events: fever ≥37.8 ºC; urinary tract infection (UTI) or sepsis (standardized definition). We will also evaluate the predictive factors of infectious complications

ELIGIBILITY:
Inclusion Criteria:

* Signature of the consent term;
* Agreement with the study follow-up protocol;
* Indication of biopsy due to increased PSA (> 2.5), abnormal rectal touch or patients under active surveillance protocol

Exclusion Criteria:

* Existence of cognitive deficit that impedes the reading and comprehension of the EHIC;
* Allergy to ciprofloxacin or iodine

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Infectious complications | 1 week
  compare the infectious outcomes of intrarectal povidone-iodine cleansing plus formalin disinfection of needle tip during transrectal ultrasound guided prostate biopsy

SECONDARY OUTCOMES:
evaluate predictive factors of infectious complications after prostate biopsy. | 1 week
  evaluate predictive factors of infectious complications after prostate biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Transplantes Euryclides de Jesus Zerbini, São Paulo, Brazil

REFERENCES:
- [Background] Noguchi M, Matsuoka K, Koga H, Kanetake H, Nakagawa M, Naito S. A questionnaire survey of patient preparation and techniques for prostate biopsy among urologists in the Kyushu and Okinawa regions of Japan. Int J Clin Oncol. 2006 Oct;11(5):390-5. doi: 10.1007/s10147-006-0592-3. PMID 17058137
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Zappa M, Nelen V, Kwiatkowski M, Lujan M, Maattanen L, Lilja H, Denis LJ, Recker F, Paez A, Bangma CH, Carlsson S, Puliti D, Villers A, Rebillard X, Hakama M, Stenman UH, Kujala P, Taari K, Aus G, Huber A, van der Kwast TH, van Schaik RH, de Koning HJ, Moss SM, Auvinen A; ERSPC Investigators. Screening and prostate cancer mortality: results of the European Randomised Study of Screening for Prostate Cancer (ERSPC) at 13 years of follow-up. Lancet. 2014 Dec 6;384(9959):2027-35. doi: 10.1016/S0140-6736(14)60525-0. Epub 2014 Aug 6. PMID 25108889
- [Background] Zaytoun OM, Vargo EH, Rajan R, Berglund R, Gordon S, Jones JS. Emergence of fluoroquinolone-resistant Escherichia coli as cause of postprostate biopsy infection: implications for prophylaxis and treatment. Urology. 2011 May;77(5):1035-41. doi: 10.1016/j.urology.2010.12.067. Epub 2011 Mar 21. PMID 21420152
- [Background] Djavan B, Waldert M, Zlotta A, Dobronski P, Seitz C, Remzi M, Borkowski A, Schulman C, Marberger M. Safety and morbidity of first and repeat transrectal ultrasound guided prostate needle biopsies: results of a prospective European prostate cancer detection study. J Urol. 2001 Sep;166(3):856-60. PMID 11490233
- [Background] Zani EL, Clark OA, Rodrigues Netto N Jr. Antibiotic prophylaxis for transrectal prostate biopsy. Cochrane Database Syst Rev. 2011 May 11;2011(5):CD006576. doi: 10.1002/14651858.CD006576.pub2. PMID 21563156
- [Background] Lindstedt S, Lindstrom U, Ljunggren E, Wullt B, Grabe M. Single-dose antibiotic prophylaxis in core prostate biopsy: Impact of timing and identification of risk factors. Eur Urol. 2006 Oct;50(4):832-7. doi: 10.1016/j.eururo.2006.05.003. Epub 2006 May 16. PMID 16750292
- [Background] Lee SJ. Infection after transrectal ultrasound-guided prostate biopsy. Korean J Urol. 2015 May;56(5):346-50. doi: 10.4111/kju.2015.56.5.346. Epub 2015 Apr 6. PMID 25964834
- [Background] Carignan A, Roussy JF, Lapointe V, Valiquette L, Sabbagh R, Pepin J. Increasing risk of infectious complications after transrectal ultrasound-guided prostate biopsies: time to reassess antimicrobial prophylaxis? Eur Urol. 2012 Sep;62(3):453-9. doi: 10.1016/j.eururo.2012.04.044. Epub 2012 May 3. PMID 22575912
- [Background] Feliciano J, Teper E, Ferrandino M, Macchia RJ, Blank W, Grunberger I, Colon I. The incidence of fluoroquinolone resistant infections after prostate biopsy--are fluoroquinolones still effective prophylaxis? J Urol. 2008 Mar;179(3):952-5; discussion 955. doi: 10.1016/j.juro.2007.10.071. Epub 2008 Jan 22. PMID 18207185
- [Background] Liss MA, Chang A, Santos R, Nakama-Peeples A, Peterson EM, Osann K, Billimek J, Szabo RJ, Dash A. Prevalence and significance of fluoroquinolone resistant Escherichia coli in patients undergoing transrectal ultrasound guided prostate needle biopsy. J Urol. 2011 Apr;185(4):1283-8. doi: 10.1016/j.juro.2010.11.088. Epub 2011 Feb 22. PMID 21334021
- [Background] Duplessis CA, Bavaro M, Simons MP, Marguet C, Santomauro M, Auge B, Collard DA, Fierer J, Lesperance J. Rectal cultures before transrectal ultrasound-guided prostate biopsy reduce post-prostatic biopsy infection rates. Urology. 2012 Mar;79(3):556-61. doi: 10.1016/j.urology.2011.09.057. PMID 22386395
- [Background] Fahmy A, Rhashad H, Mohi M, Elabbadie A, Kotb A. Optimizing prophylactic antibiotic regimen in patients admitted for transrectal ultrasound-guided prostate biopsies: A prospective randomized study. Prostate Int. 2016 Sep;4(3):113-7. doi: 10.1016/j.prnil.2016.06.001. Epub 2016 Jul 1. PMID 27689069
- [Background] Steensels D, Slabbaert K, De Wever L, Vermeersch P, Van Poppel H, Verhaegen J. Fluoroquinolone-resistant E. coli in intestinal flora of patients undergoing transrectal ultrasound-guided prostate biopsy--should we reassess our practices for antibiotic prophylaxis? Clin Microbiol Infect. 2012 Jun;18(6):575-81. doi: 10.1111/j.1469-0691.2011.03638.x. Epub 2011 Sep 29. PMID 21958149
- [Background] Taylor AK, Zembower TR, Nadler RB, Scheetz MH, Cashy JP, Bowen D, Murphy AB, Dielubanza E, Schaeffer AJ. Targeted antimicrobial prophylaxis using rectal swab cultures in men undergoing transrectal ultrasound guided prostate biopsy is associated with reduced incidence of postoperative infectious complications and cost of care. J Urol. 2012 Apr;187(4):1275-9. doi: 10.1016/j.juro.2011.11.115. Epub 2012 Feb 16. PMID 22341272
- [Background] Jeon SS, Woo SH, Hyun JH, Choi HY, Chai SE. Bisacodyl rectal preparation can decrease infectious complications of transrectal ultrasound-guided prostate biopsy. Urology. 2003 Sep;62(3):461-6. doi: 10.1016/s0090-4295(03)00470-9. PMID 12946747
- [Background] Carey JM, Korman HJ. Transrectal ultrasound guided biopsy of the prostate. Do enemas decrease clinically significant complications? J Urol. 2001 Jul;166(1):82-5. PMID 11435829
- [Background] Zaytoun OM, Anil T, Moussa AS, Jianbo L, Fareed K, Jones JS. Morbidity of prostate biopsy after simplified versus complex preparation protocols: assessment of risk factors. Urology. 2011 Apr;77(4):910-4. doi: 10.1016/j.urology.2010.12.033. Epub 2011 Feb 12. PMID 21316093
- [Background] Abughosh Z, Margolick J, Goldenberg SL, Taylor SA, Afshar K, Bell R, Lange D, Bowie WR, Roscoe D, Machan L, Black PC. A prospective randomized trial of povidone-iodine prophylactic cleansing of the rectum before transrectal ultrasound guided prostate biopsy. J Urol. 2013 Apr;189(4):1326-31. doi: 10.1016/j.juro.2012.09.121. Epub 2012 Oct 2. PMID 23041343
- [Background] Singla N, Walker J, Woldu SL, Passoni NM, de la Fuente K, Roehrborn CG. Formalin disinfection of prostate biopsy needles may reduce post-biopsy infectious complications. Prostate Cancer Prostatic Dis. 2017 Jun;20(2):216-220. doi: 10.1038/pcan.2016.70. Epub 2017 Jan 24. PMID 28117384
- [Background] Valverde A, Msika S, Kianmanesh R, Hay JM, Couchard AC, Flamant Y, Fingerhut A, Fagniez PL; French Associations for Surgical Research. Povidone-iodine vs sodium hypochlorite enema for mechanical preparation before elective open colonic or rectal resection with primary anastomosis: a multicenter randomized controlled trial. Arch Surg. 2006 Dec;141(12):1168-74; discussion 1175. doi: 10.1001/archsurg.141.12.1168. PMID 17178958
- [Background] Park DS, Oh JJ, Lee JH, Jang WK, Hong YK, Hong SK. Simple use of the suppository type povidone-iodine can prevent infectious complications in transrectal ultrasound-guided prostate biopsy. Adv Urol. 2009;2009:750598. doi: 10.1155/2009/750598. Epub 2009 Apr 23. PMID 19404480
- [Background] Goh YS, Law ZW, Tiong HY. Re: A prospective randomized trial of povidone-iodine prophylactic cleansing of the rectum before transrectal ultrasound guided prostate biopsy: Z. AbuGhosh, J. Margolick, S. L. Goldenberg, S. A. Taylor, K. Afshar, R. Bell, D. Lange, W. R. Bowie, D. Roscoe, L. Machan and P. C. Black J Urol 2013; 189: 1326-1331. J Urol. 2013 Dec;190(6):2309-10. doi: 10.1016/j.juro.2013.07.010. Epub 2013 Sep 17. No abstract available. PMID 24050910
- [Background] Zembower TR, Maxwell KM, Nadler RB, Cashy J, Scheetz MH, Qi C, Schaeffer AJ. Evaluation of targeted antimicrobial prophylaxis for transrectal ultrasound guided prostate biopsy: a prospective cohort trial. BMC Infect Dis. 2017 Jun 7;17(1):401. doi: 10.1186/s12879-017-2470-1. PMID 28592230
- [Background] Naughton CK, Miller DC, Mager DE, Ornstein DK, Catalona WJ. A prospective randomized trial comparing 6 versus 12 prostate biopsy cores: impact on cancer detection. J Urol. 2000 Aug;164(2):388-92. PMID 10893592